CLINICAL TRIAL: NCT00098956
Title: A Phase II Study of UCN-01 in Combination With Topotecan in Patients With SCLC Who Relapsed or Progressed >= 3 Months After Completing First-Line Platinum-Based Chemotherapy
Brief Title: 7-hydroxystaurosporine and Topotecan Hydrochloride in Treating Patients With Relapsed or Progressed Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03092; NCI-2012-03092 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 6992; PHL032 (Other: Princess Margaret Hospital Phase 2 Consortium); 6992 (Other: CTEP); N01CM62203 (NIH)
Record Dates: First submitted 2004-12-08; First posted 2004-12-09 (Estimated); Results first posted 2015-09-09 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Extensive Stage Small Cell Lung Cancer; Recurrent Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Topotecan; trioctyl phosphine oxide; 7-hydroxystaurosporine

ARMS (1):
- Treatment (topotecan hydrochloride, UCN-01) (Experimental): Patients receive topotecan IV over 30 minutes on days 1-5 and UCN-01 IV over 3 hours on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients achieving CR or PR receive 2 additional courses beyond CR or PR.
  Interventions: Drug: topotecan hydrochloride; Drug: 7-hydroxystaurosporine

INTERVENTIONS:
Drug: topotecan hydrochloride — Given IV
  Other Names: hycamptamine; Hycamtin; SKF S-104864-A; TOPO
Drug: 7-hydroxystaurosporine — Given IV
  Other Names: UCN-01

SUMMARY:
This phase II trial is studying how well giving UCN-01 together with topotecan works in treating patients with small cell lung cancer that relapsed or progressed after previous chemotherapy. Drugs used in chemotherapy, such as topotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. UCN-01 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It may also increase the effectiveness of topotecan by making tumor cells more sensitive to the drug. Giving UCN-01 together with topotecan may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the anti tumour activity of UCN-01 in combination with topotecan in patients with SCLC who relapsed or progressed >= 3 months after completing first-line platinum-based chemotherapy (patient with sensitive disease) using objective response rates (complete and partial).

SECONDARY OBJECTIVES:

I. To determine the anti tumour activity of UCN-01 in combination with topotecan with regards to stable disease rate, median and overall survival rates as well as to determine the safety and tolerability of this combination.

OUTLINE: This is a multicenter study.

Patients receive topotecan IV over 30 minutes on days 1-5 and UCN-01 IV over 3 hours on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients achieving complete response (CR) or partial response (PR) receive 2 additional courses beyond CR or PR.

Patients are followed for survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed extensive stage small cell lung cancer that is incurable but amenable to treatment with chemotherapy
* Patients must have measurable disease as defined by the Response Evaluation Criteria in Solid Tumours (RECIST); they must have either measurable disease outside the field or progression post radiation therapy
* Patient must have received ONLY first-line platinum-based chemotherapy and relapsed or progressed >= 3 months post completion of therapy (patients with chemo-sensitive disease)
* Patient must have completed any prior chemotherapy at least 3 months before study entry, have completed surgery or radiotherapy at least 4 weeks before study entry and must have recovered from the toxic effects from any prior therapy; patient must not have had more than 40% of their bone marrow radiated
* ECOG performance status =< 2 (Karnofsky >= 60%)
* Leucocytes >= 3 x 10^9/L OR
* ANC >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Total serum bilirubin =< 1.5 x UNL
* AST/ALT =< 3 x UNL (=< 5 x UNL if documented liver metastases)
* Creatinine =< institutional upper limit of normal OR creatinine clearance >= 50 ml/min/1.73m^2 for patients with creatinine levels above institutional normal
* The effects of UCN-01 on the developing human fetus are unknown; for this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation; contraception should be continued at least 3 months after the last dose of UCN-01; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had prior therapy with a topoisomerase I inhibitor (topotecan or irinotecan) will be excluded
* Patients who have had other chemotherapy regimens other than first-line platinum-based chemotherapy will be excluded
* Patients may not be receiving any other investigational agents
* Patients may not be receiving concurrent radiation therapy while on study treatment
* Patients with uncontrolled/symptomatic CNS metastases; routine CT scans are not required to rule these out except when there is clinical suspicion of CNS disease
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to UCN-01 or other agents used in study
* Because of cardiopulmonary toxicity seen in patients on other studies, patients with a history of coronary artery disease and/or symptomatic cardiac dysfunction should be excluded
* Because UCN-01 may cause hyperglycemia, patients with insulin dependent diabetes mellitus will be excluded; patients with diet-controlled diabetes mellitus or those on oral hypoglycemic agents can be entered at the discretion of the investigator
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because UCN-01 is a serine-threonine kinase inhibitor with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with UCN-01, breastfeeding should be discontinued if the mother is treated with UCN-01; these potential risks may also apply to other agents used in this study
* Because patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with UCN-01 or other agents administered during the study; appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated
* Patients may not have had any other active malignancy in the past 5 years except for cervical carcinoma in situ and non-melanomatous skin cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2005-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glennwood Goss, Principal Investigator — Princess Margaret Hospital Phase 2 Consortium
Locations (1):
- Princess Margaret Hospital Phase 2 Consortium, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Topotecan Hydrochloride, UCN-01)
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Topotecan Hydrochloride, UCN-01)
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 7
Age, Continuous [Mean (Full Range); unit: years] | 59 [51 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 9
Region of Enrollment [Number; unit: participants]
  Canada | 19

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rates (Complete and Partial) Evaluated Using RECIST Criteria
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Objective Response (OR) = CR + PR.
Time Frame: Up to 5 years
Measure: Number; unit: participants
Arm/Group | Treatment (Topotecan Hydrochloride, UCN-01)
Number analyzed (Participants) | 19
participants | 2

2. Secondary Outcome: Stable Disease Rate Evaluated Using RECIST Criteria
Description: Per Response Evaluation Criteria In Solid Tumours Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), at least 30% decrease in the sum of the longest diameter of target lesions; Objective Response (OR) = CR + PR.
Time Frame: Up to 5 years
Measure: Number; unit: participants
Arm/Group | Treatment (Topotecan Hydrochloride, UCN-01)
Number analyzed (Participants) | 19
participants | 9

3. Secondary Outcome: Duration of Responses
Time Frame: From the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, assessed up to 5 years
Population: Data were not collected
Arm/Group | Treatment (Topotecan Hydrochloride, UCN-01)
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression-free Survival
Time Frame: From the date of enrollment to progression, death or last contact, or last tumor assessment before the start of further anti-tumor therapy, assessed up to 5 years
Population: Data were not collected
Arm/Group | Treatment (Topotecan Hydrochloride, UCN-01)
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival
Time Frame: From the date of enrollment to death or last contact, assessed up to 5 years
Population: Data were not collected
Arm/Group | Treatment (Topotecan Hydrochloride, UCN-01)
Number analyzed (Participants) | 0

6. Secondary Outcome: Adverse Events, Graded Using the CTCAE Version 3.0
Time Frame: Up to 5 years
Measure: Number; unit: types of grade 3 / 4 toxicities reported
Arm/Group | Treatment (Topotecan Hydrochloride, UCN-01)
Number analyzed (Participants) | 17
types of grade 3 / 4 toxicities reported | 7

ADVERSE EVENTS:
Arm/Group | Treatment (Topotecan Hydrochloride, UCN-01)
Serious Adverse Events (participants affected / at risk) | 3/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Topotecan Hydrochloride, UCN-01) (N=19)
Death NOS (General disorders) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 1 (1)
Cardiac disorder other (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Topotecan Hydrochloride, UCN-01) (N=19)
Neutrophil count decreased (Investigations) | 13 (13)
White blood cell decreased (Investigations) | 14 (14)
Platelet count decreased (Investigations) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less